CLINICAL TRIAL: NCT00660920
Title: A Phase 1 Dose Escalation Trial to Determine the Safety, Tolerability and Maximum Tolerated Dose of Oral AP24534 in Patients With Refractory or Advanced Chronic Myelogenous Leukemia and Other Hematologic Malignancies
Brief Title: Safety Study of AP24534 to Treat Chronic Myelogenous Leukemia (CML) and Other Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP24534-07-101
Expanded Access: NCT01592136 (Approved for marketing)
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-02

CONDITIONS: Chronic Myelogenous Leukemia; Hematologic Malignancies
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hematologic Neoplasms | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ponatnib (Experimental): Comparison of different dosages of ponatinib given orally once per day.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Comparison of different dosages of drug given orally once per day.
  Other Names: AP24534; Iclusig

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose or a recommended dose of oral AP24534 in a defined schedule in patients with refractory or advanced chronic myelogenous leukemia and other refractory hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 years old
* Diagnosed hematologic malignancy (other than lymphoma) that has relapsed or is refractory to standard care or for which no standard care is available or acceptable
* Able to give written informed consent
* ECOG performance status ≤ 2
* BSA ≥ 1.5 m² (first cohort only)
* Minimum life expectancy of 3 months or more
* Adequate renal function defined as serum creatinine <1.5× upper limit of normal (ULN) for institution
* Adequate hepatic function (defined as: Total bilirubin <1.5 × ULN for institution; ALT and AST <2.5 × ULN for institution [<5 X ULN if liver involvement with leukemia]; Prothrombin time <1.5 × ULN)
* Ability to comply with study procedures in the Investigator's opinion
* Adequate cardiac function defined as ejection fraction (EF) >40% by any method of the investigator's choice
* Normal QTcF interval on screening ECG evaluation, defined as QTcF of <450 ms.
* For females of childbearing potential, a negative pregnancy test must be documented prior to enrollment
* Female patients who are of childbearing potential must agree to use an effective form of contraception with their sexual partners throughout participation in this study

Exclusion Criteria:

* Have had cytotoxic chemotherapy or radiotherapy within 21 days prior to entering the study, or those who have not recovered from adverse events due to agents administered more than 28 days earlier with the exception of alopecia
* Received any other investigational agents or have received an investigational agent within 14 days of starting ponatinib
* Malabsorption syndrome or other illness which could affect oral absorption
* Significant uncontrolled cardiac disease
* Patients taking medicinal products that are known to be associated with prolongation of the QT interval on the electrocardiogram.
* Uncontrolled hypertension (Diastolic BP >100 mmHg; Systolic >150 mmHg)
* Uncontrolled intercurrent illness
* Pregnant
* Known infection with HIV
* Autologous or allogeneic stem cell transplant < 3 months prior to enrollment; any evidence of ongoing graft versus host disease (GVHD), or GVHD requiring immunosuppressive therapy
* Another primary malignancy within the past 3 years
* Any condition or illness which, in the opinion of the investigator, would compromise patient safety or interfere with the evaluation of the safety of the drug
* Patients taking medicinal products that are known to be associated with prolongation of the QT interval on the electrocardiogram
* Major surgery (with the exception of intravenous catheter placement or bone marrow biopsy) within 14 days prior to initiating ponatinib therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Determine Maximum Tolerated Dose (MTD) or Recommended dose | Up to
  Determine MTD dose or a recommended dose of oral ponatinib in a defined schedule (QD) in patients with refractory or advanced chronic myelogenous leukemia and other refractory hematologic malignancies.

SECONDARY OUTCOMES:
To examine the safety of AP24534 in patients with resistant/refractory hematologic malignancies | Up to 7 years
To describe the anti-tumor activity of AP24534 in patients with refractory hematologic malignancies | Up to 7 years
To examine the pharmacokinetics of AP24534 | Up to 2 cycles (1 cycle = 28 days)
To examine pharmacodynamic activity of AP24534 in CML and Ph + ALL patients | Up to 7 years
To describe potential pharmacogenomic markers of AP24534 anti-tumor activity | Up to 7 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - ARIAD Investigational Site #075, San Francisco, California
  - ARIAD Investigational Site #011, Ann Arbor, Michigan
  - ARIAD Investigational Site #048, Portland, Oregon
  - ARIAD Investigational Site #076, Nashville, Tennessee
  - ARIAD Investigational Site #005, Houston, Texas

REFERENCES:
- [Derived] Hanley MJ, Diderichsen PM, Narasimhan N, Srivastava S, Gupta N, Venkatakrishnan K. Population Pharmacokinetics of Ponatinib in Healthy Adult Volunteers and Patients With Hematologic Malignancies and Model-Informed Dose Selection for Pediatric Development. J Clin Pharmacol. 2022 Apr;62(4):555-567. doi: 10.1002/jcph.1990. Epub 2021 Dec 16. PMID 34699069
- [Derived] Cortes JE, Kantarjian H, Shah NP, Bixby D, Mauro MJ, Flinn I, O'Hare T, Hu S, Narasimhan NI, Rivera VM, Clackson T, Turner CD, Haluska FG, Druker BJ, Deininger MW, Talpaz M. Ponatinib in refractory Philadelphia chromosome-positive leukemias. N Engl J Med. 2012 Nov 29;367(22):2075-88. doi: 10.1056/NEJMoa1205127. PMID 23190221